CLINICAL TRIAL: NCT01217593
Title: A Comparison Of Ultrasound and Predetermined Distance Techniques For Paravertebral Space Localization In Breast Surgery: A Randomized Prospective Trial
Brief Title: Ultrasound vs. Predetermined Distance Techniques for Paravertebral Nerve Block in Patients Having Breast Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ochsner Health System (Other)
Responsible Party: Principal Investigator, Kristie Osteen, Director of Perioperative Anesthesia, Ochsner Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2010.116.C; PI-Osteen (Other: Ochnser Clinic Foundation Institutional Review Board)
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Mastectomy; Breast Neoplasms
Keywords: mastectomy; breast cancer; breast surgery
MeSH Terms: conditions — Breast Neoplasms | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ultrasound (Experimental): Ultrasound guidance will be used for paravertebral space localization when performing paravertebral blocks on females 25-85 having unilateral mastectomy.
  Interventions: Procedure: ultrasound
- predetermined distance (Active Comparator): The predetermined distance technique will be used for paravertebral space localization when performing paravertebral blocks on females 25-85 having unilateral mastectomy.
  Interventions: Procedure: predetermined distance

INTERVENTIONS:
Procedure: ultrasound — Ultrasound guidance will be used for paravertebral space localization when performing paravertebral blocks on females 25-85 having unilateral mastectomy.
  Arms: ultrasound
Procedure: predetermined distance — The predetermined distance technique will be used for paravertebral space localization when performing paravertebral blocks on females 25-85 having unilateral mastectomy.
  Arms: predetermined distance

SUMMARY:
The purpose of this study is to compare ultrasound and predetermined distance techniques for finding the paravertebral space to inject the local anesthetic (numbing medicine) when you are given anesthesia for surgery. The paravertebral space is located on either side of the spinal cord and contains the nerves that provide sensation to the chest wall. The predetermined distance technique is a series of measurements taken to determine the location of the paravertebral space where the local anesthetic is injected. The ultrasound technique uses direct visualization of the local anesthetic being placed in the paravertebral space. This type of anesthesia has many benefits including decreasing your pain after breast surgery.

ELIGIBILITY:
Inclusion Criteria:

* Females age 25 - 85
* ASA Physical status I-III
* Scheduled for primary mastectomy
* Ability to give informed consent

Exclusion Criteria:

* Allergy to:

Local anesthetics Fentanyl Hydromorphone Propofol Midazolam

* Patient refusal
* Infection at the injection site
* Peripheral Neuropathy
* Bilateral breast surgery
* Prior thoracic surgery on surgical side
* Severe spinal deformity
* Coagulopathy

Ages: 25 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Visual analog scores(VAS)for pain and perioperative opioid requirements | 24 hours
  The VAS scores and the opioid consumption will be compared between the ultrasound group and the predetermined distance technique group.

SECONDARY OUTCOMES:
time, incidence of adverse events and patient satisfaction | 24 hours
  The secondary objectives will be 1) time taken to locate the paravertebral space and inject local anesthetic 2) time from injection of local anesthetic to adequate sensory block 3) incidence of adverse events including pneumothorax, high spinal, epidural spread, direct nerve damage, paresthesias, vascular puncture, patient discomfort, respiratory depression, hypoxemia, and prolonged sensory blockade and 4) patient satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Kristie Osteen, MD, Principal Investigator — Ochsner Health System
Locations (1):
- Ochsner Clinic Foundation, New Orleans, Louisiana, United States

REFERENCES:
- [Background] la Grange P, Foster PA, Pretorius LK. Application of the Doppler ultrasound bloodflow detector in supraclavicular brachial plexus block. Br J Anaesth. 1978 Sep;50(9):965-7. doi: 10.1093/bja/50.9.965. PMID 708565
- [Result] Marhofer P, Schrogendorfer K, Koinig H, Kapral S, Weinstabl C, Mayer N. Ultrasonographic guidance improves sensory block and onset time of three-in-one blocks. Anesth Analg. 1997 Oct;85(4):854-7. doi: 10.1097/00000539-199710000-00026. PMID 9322469
- [Result] Domingo-Triado V, Selfa S, Martinez F, Sanchez-Contreras D, Reche M, Tecles J, Crespo MT, Palanca JM, Moro B. Ultrasound guidance for lateral midfemoral sciatic nerve block: a prospective, comparative, randomized study. Anesth Analg. 2007 May;104(5):1270-4, tables of contents. doi: 10.1213/01.ane.0000221469.24319.49. PMID 17456685
- [Result] Willschke H, Marhofer P, Bosenberg A, Johnston S, Wanzel O, Cox SG, Sitzwohl C, Kapral S. Ultrasonography for ilioinguinal/iliohypogastric nerve blocks in children. Br J Anaesth. 2005 Aug;95(2):226-30. doi: 10.1093/bja/aei157. Epub 2005 May 27. PMID 15923270
- [Result] Oberndorfer U, Marhofer P, Bosenberg A, Willschke H, Felfernig M, Weintraud M, Kapral S, Kettner SC. Ultrasonographic guidance for sciatic and femoral nerve blocks in children. Br J Anaesth. 2007 Jun;98(6):797-801. doi: 10.1093/bja/aem092. Epub 2007 Apr 21. PMID 17449890
- [Result] Deegan CA, Murray D, Doran P, Ecimovic P, Moriarty DC, Buggy DJ. Effect of anaesthetic technique on oestrogen receptor-negative breast cancer cell function in vitro. Br J Anaesth. 2009 Nov;103(5):685-90. doi: 10.1093/bja/aep261. Epub 2009 Sep 22. PMID 19776028
- [Result] Boughey JC, Goravanchi F, Parris RN, Kee SS, Kowalski AM, Frenzel JC, Bedrosian I, Meric-Bernstam F, Hunt KK, Ames FC, Kuerer HM, Lucci A. Prospective randomized trial of paravertebral block for patients undergoing breast cancer surgery. Am J Surg. 2009 Nov;198(5):720-5. doi: 10.1016/j.amjsurg.2008.11.043. Epub 2009 May 9. PMID 19427625
- [Result] Goldfarb Y, Ben-Eliyahu S. Surgery as a risk factor for breast cancer recurrence and metastasis: mediating mechanisms and clinical prophylactic approaches. Breast Dis. 2006-2007;26:99-114. doi: 10.3233/bd-2007-26109. PMID 17473369
- [Result] Coveney E, Weltz CR, Greengrass R, Iglehart JD, Leight GS, Steele SM, Lyerly HK. Use of paravertebral block anesthesia in the surgical management of breast cancer: experience in 156 cases. Ann Surg. 1998 Apr;227(4):496-501. doi: 10.1097/00000658-199804000-00008. PMID 9563536